CLINICAL TRIAL: NCT01099033
Title: The Biologic Basis of Hernia Formation
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 201104031
Record Dates: First submitted 2010-04-02; First posted 2010-04-06 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Hiatal Hernia; Paraesophageal Hernia
Keywords: hiatal hernia; paraesophageal hernia; biologic mesh; MMPs; Hiatal/Paraesophageal hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — small tissue biopsies of gastrohepatic, gastrophrenic, and phrenoesophageal ligaments
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hiatal/Paraesophageal hernia patients: patients with hiatal or paraesophageal hernias
- control group: patients without hiatal or paraesophageal hernias who are undergoing crural dissection for heller myotomy, or who are undergoing gastric bypass surgery

SUMMARY:
The study will examine potential biological and genetic mechanisms leading to hiatal and paraesophageal hernia formation in predisposed individuals. It is expected that these patients will have defects in the normal production and maturation of collagen and other connective tissue proteins, thus leading to weakness in the diaphragm that may allow for spontaneous herniation. Comparison of tissue and blood samples from these patients (study group) will be made to those from individuals undergoing lower esophageal surgery who have not developed a concurrent hernia (i.e. esophageal myotomy for achalasia and laparoscopic gastric bypass or laparoscopic adjustable gastric banding for morbid obesity - control group).

DETAILED DESCRIPTION:
Diaphragmatic herniation is a common medical problem characterized by protrusion of the abdominal viscera directly through (95% of cases), or adjacent to (5% of cases), the esophageal hiatus. Individuals suffering from these so-called hiatal and paraesophageal hernias experience symptoms such as regurgitation, heartburn, early satiety, and in extreme cases, respiratory compromise or visceral strangulation and ischemia. Unless the hernia is small, these symptoms are generally refractory to medical management and require surgical correction, with approximately 40,000 antireflux surgeries being performed each year in the United States. The hernia repair procedure, which may be performed in either a laparoscopic or open fashion, involves reduction of the intrathoracic viscera back into the abdominal cavity and closure of the diaphragmatic defect. Generally, this closure of the hernia can be accomplished primarily, using nonabsorbable suture to approximate the edges of the defect. Unfortunately, the recurrence rate for this type of repair is unacceptably high and ranges from 10-40%. Furthermore, in the instance of a particularly large hernia, the edges of the defect may be too far apart to be primarily brought together, necessitating the use of other strategies such as relaxing incisions or patches to bridge the gap. Although the precise recurrence rates of these complex repairs is not clear, it is expected that they are even higher that for those diaphragmatic hernias that can be closed primarily.

The genetic and biologic factors that predispose individuals to forming hernias are not well understood. Several smaller series have suggested that ventral and inguinal hernia formation may be due to weakness of the abdominal wall, possibly secondary to defects in collagen deposition and metabolism. Certain studies have shown higher ratios of Type III collagen (immature) to Type I collagen (mature), at both the protein and mRNA level, in patients with abdominal hernias as compared to those without. Furthermore, other reports indicate that these differences in the levels of mature collagen might be due to underlying differences ion the expression of certain matrix metalloproteinase (MMPs), which are largely responsible for collagen remodeling. MMPs -1, -2, -3, -9, and -13 have been shown to be upregulated in connective tissue injury, and alterations in both MMP-2 and fibrillar collagen can interfere with normal wound healing. Furthermore, Bellon et. al. have shown an overexpression of MMP-2 in fibroblasts in patients with direct inguinal hernias, and Zheng's group detected MMP-13 overexpression in tissue samples from patients with recurrent inguinal hernias. So far, no studies have addressed the role of collagen deposition and MMPs in the formation of hiatal and paraesophageal hernias. Preliminary work at our institution has, however, shown a greater than 50% reduction in the elastin content of the phrenoesophageal and gastrohepatic ligaments ("PEL" and "GHL", respectively) of those patients with a hiatal hernia compared to those without herniation. Additionally, the elastic fibers in the PEL and GHL frequently displayed fragmentation and distortion despite the lack of a visible inflammatory response. (J.A. Curci and N.J. Soper, unpublished results) Nevertheless, neither our early work, nor any of the studies from outside institutions have looked at ways of screening patients (i.e. via blood sampling) to detect those at a higher risk for such hernia occurrence. Currently, new MMP-inhibitory drugs are being studied as methods to potentially block or slow the development of other MMP-dependent conditions such as abdominal aortic aneurysm (AAA). Along these lines, if patients with a genetic/biologic predisposition to hernia formation could be readily identified, then this presents a potential point of medical intervention in preventing future hernia development.

Research procedures:

Patients to be enrolled in the study will be standard referrals to our group from primary care physicians or other specialists who feel that surgical correction of a diaphragmatic hernia or achalasia is necessary. Additionally, patients referred to our practice for weight reduction surgery will also be considered eligible for enrollment.

Consent to participate in the study will occur at the time of consent to the surgical procedure and will be obtained by the PI and other attending surgeons within the minimally invasive surgery group. This will occur in the surgeon's office/clinic, or in the hospital if the patient is an in-house consult, several days to weeks prior to the scheduled surgery.

Following the informed consent process, patients will be appropriately placed in either the study or control group. At the time of surgery (hernia repair, bariatric procedure, or esophageal myotomy), a 30 ml venous blood sample will be drawn and stored for later testing and analysis. The appropriate standard surgical procedure will then be performed as per surgical attending judgment, however, during the operation, a small (approximately 1 cm2) piece of tissue will be excised from each of 3 anatomic sites: 1) the left diaphragmatic crus, 2) the PEL, and 3) the GHL. After removal from the abdomen, these tissue samples will be divided into 2 pieces to be set aside for further testing at a later time.

This excised samples represent a minute amount of tissue when compared to the overall size of the diaphragmatic crura and surrounding ligamentous attachments, and their removal is not be expected to cause any foreseeable problem for the patient. In fact, hiatal hernia repair often necessitates dissection of much larger crural and connective tissue pieces than this in order to obtain complete reduction of the abdominal viscera out of the chest and subsequent closure of the hernia defect. Following removal of these small tissue samples, the hernia repair, esophageal myotomy, or gastric bypass/banding will then be completed in a standard fashion.

Inclusion Criteria: Any patient undergoing paraesophageal hernia repair, esophageal myotomy, laparoscopic gastric bypass, or laparoscopic adjustable gastric banding.

Exclusion Criteria: Pregnant females, minors, prisoners

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing paraesophageal hernia repair, esophageal myotomy, laparoscopic gastric bypass, or laparoscopic adjustable gastric banding.

Exclusion Criteria:

* Pregnant females, minors, prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to be enrolled in the study will be standard referrals to our group from primary care physicians or other specialists who feel that surgical correction of a diaphragmatic hernia or achalasia is necessary. Additionally, patients referred to our practice for weight reduction surgery will also be considered eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2007-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent D Matthews, MD, Principal Investigator — Washington University School of Medicine; Corey Deeken, PhD, Study Director — Washington University School of Medicine; Peggy Frisella, RN, Study Chair — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Jansen PL, Mertens Pr Pr, Klinge U, Schumpelick V. The biology of hernia formation. Surgery. 2004 Jul;136(1):1-4. doi: 10.1016/j.surg.2004.01.004. No abstract available. PMID 15232531
- [Background] Klinge U, Si ZY, Zheng H, Schumpelick V, Bhardwaj RS, Klosterhalfen B. Abnormal collagen I to III distribution in the skin of patients with incisional hernia. Eur Surg Res. 2000;32(1):43-8. doi: 10.1159/000008740. PMID 10720845